CLINICAL TRIAL: NCT06592261
Title: Human Models of Selective Insulin Resistance: Graded Insulin Suppression Test (GIST) Pilot & Feasibility Study
Brief Title: Graded Insulin Suppression Test P&F
Acronym: GIST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Pisa (Other)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAAV2481; 3P30DK063608-21 (NIH); K12DK133995 (NIH); K23DK140614 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Insulin Resistance; Hyperinsulinemia; Obesity; Healthy
Keywords: Insulin resistance; Hyperinsulinemia; Type 2 diabetes; Obesity
MeSH Terms: conditions — Insulin Resistance; Hyperinsulinism; Obesity; Diabetes Mellitus, Type 2 | interventions — Insulin; Octreotide; Glucose; Water; Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Reference (healthy control) group (Experimental): Healthy volunteers with body mass index of 18-25 kg/m2, fasting serum insulin < 10 mU/L, hemoglobin A1c < 5.7%, and fasting plasma glucose < 100 mg/dL
  Interventions: Drug: Insulin regular, 2.0-3.2 mU/m2/min (euinsulinemia); Drug: Insulin regular, 32 mU/m2/min (hyperinsulinemia); Drug: Octreotide Acetate, 6-45 ng/kg/min; Drug: Dextrose 20 % in Water; Drug: Glucagon, 0-0.5 ng/kg/min
- Euinsulinemic group (Experimental): Volunteers with body mass index of 30-45 kg/m2, fasting serum insulin < 10 mU/L, hemoglobin A1c < 5.7%, and fasting plasma glucose < 100 mg/dL
  Interventions: Drug: Insulin regular, 2.0-3.2 mU/m2/min (euinsulinemia); Drug: Insulin regular, 32 mU/m2/min (hyperinsulinemia); Drug: Octreotide Acetate, 6-45 ng/kg/min; Drug: Dextrose 20 % in Water; Drug: Glucagon, 0-0.5 ng/kg/min
- Hyperinsulinemic group (Experimental): Volunteers with body mass index of 30-45 kg/m2, fasting serum insulin >= 13 mU/L, hemoglobin A1c < 5.7%, and fasting plasma glucose < 100 mg/dL
  Interventions: Drug: Insulin regular, 2.0-3.2 mU/m2/min (euinsulinemia); Drug: Insulin regular, 32 mU/m2/min (hyperinsulinemia); Drug: Octreotide Acetate, 6-45 ng/kg/min; Drug: Dextrose 20 % in Water; Drug: Glucagon, 0-0.5 ng/kg/min

INTERVENTIONS:
Drug: Insulin regular, 2.0-3.2 mU/m2/min (euinsulinemia) — Insulin infusion to recapitulate euinsulinemia (normal basal insulin)
Drug: Insulin regular, 32 mU/m2/min (hyperinsulinemia) — Insulin infusion to induce hyperinsulinemia for assessment of insulin sensitivity
Drug: Octreotide Acetate, 6-45 ng/kg/min — Suppression of endogenous insulin secretion
Drug: Dextrose 20 % in Water — Production of steady-state plasma glucose (SSPG) reflective of insulin sensitivity at hyperinsulinemia
Drug: Glucagon, 0-0.5 ng/kg/min — Replacement of endogenous glucagon suppressed by octreotide. (Use is optional at the PI's discretion.)

SUMMARY:
The goal of this study is to learn about how the hormone insulin controls blood sugar in a variety of people. The main question it aims to answer is about how much insulin the body actually needs to maintain a normal blood sugar level. Participants will be asked to come in for a one-day study visit in which they will undergo a "graded insulin suppression test" ("GIST"). The GIST involves intravenous (into the vein) infusions of octreotide, a medication that turns off the body's own production of insulin, as well as replacement of insulin at two different levels (low and high), with or without replacement of glucagon, and glucose (sugar). The study investigators will check blood sugar levels every few minutes during the procedure to determine the effect of the two different insulin levels. This study will evaluate the GIST in both healthy volunteers and those at higher risk for type 2 diabetes.

DETAILED DESCRIPTION:
This study aims to determine to what extent the hyperinsulinemia commonly associated with insulin resistance (IR) in those at risk for type 2 diabetes (T2D) is a primary phenomenon, rather than merely a secondary, compensatory response to IR. The hypothesis is that some people with obesity and hyperinsulinemia exhibit a primary, non-compensatory hyperinsulinemia that may foment IR and its dysmetabolic sequelae. If this were the case, lowering insulin levels should not result in a proportional rise in blood glucose as might be expected if the hyperinsulinemia truly were purely compensatory. This hypothesis has been difficult to prove, however, because of the tight feedback mechanism between blood glucose and insulin secretion; under normal circumstances insulin secretion declines only alongside blood glucose. As such, an attempt to lower insulin levels independently of blood glucose will raise blood glucose and trigger further insulin secretion, negating the purpose of the experiment. In order to circumvent this feedback regulation of glucose-stimulated insulin secretion, this study will adapt the existing insulin suppression test (IST) technique, which employs the somatostatin receptor ligand octreotide to suppress endogenous insulin secretion and then replaces insulin and dextrose exogenously as a measure of insulin action. In addition to employing the current standard hyperinsulinemic IST protocol to assess insulin sensitivity, this study will introduce a preceding, euinsulinemic step, in which insulin is lowered toward a healthy fasting serum insulin while assessing the resultant steady-state glucose, potentially with replacement of basal glucagon. The primary endpoints in this study are the steady-state plasma glucose and serum insulin levels during low- and high-dose insulin infusions meant to induce euinsulinemia and hyperinsulinemia, respectively. The study investigators will carefully monitor plasma glucose levels every 5-15 min, drawing from an indwelling peripheral IV catheter and performing the analysis using a dedicated bedside glucose analyzer. These glucose values will be used to detect and arrest any trends toward hypo or hyperglycemia and will also serve as the readout of the primary outcome - the euinsulinemic steady-state glucose (E-SSG) and hyperinsulinemic steady-state glucose (H-SSG). Serum insulin, C-peptide, growth hormone, and glucagon levels will be measured periodically during the procedure, but these results will not be available until several days later.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18-25 and 30-45 kg/m2
* Able to understand written and spoken English and/or Spanish
* Fasting euinsulinemia (fasting serum insulin of 4-10 μU/mL) for reference group or hyperinsulinemia (fasting serum insulin ≥ 13 μU/mL) for hyperinsulinemic group on screening labs
* Written informed consent (in English or Spanish) and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

* Unable to provide informed consent in English or Spanish
* Unwillingness to use only bedpan or urinal to void or to refrain from non-emergent mobile device use during the GIST
* Documented weight loss of ≥ 5% of baseline within the previous 6 months
* Systolic blood pressure < 90 mm Hg or > 160 mm Hg, and/or
* Diastolic blood pressure < 60 mm Hg or > 100 mm Hg
* Abnormal resting heart rate: < 60 or ≥ 110 bpm
* Sinus brady or tachycardia that has been worked up and considered benign by the recruit's personal physician may be permitted at the PI's discretion
* Abnormal screening electrocardiogram (or if on file, performed within previous 90 d):

  * Non-sinus rhythm
  * Heart conduction blocks
  * Previously unknown ischaemic changes that persist on repeat EKG:
  * ST elevations
  * T-wave inversions in a vascular distribution
* Hemoglobin A1c ≥ 5.7%, and/or
* Fasting plasma glucose ≥ 100 mg/dL
* Positive qualitative β-hCG (i.e., pregnancy test) in women of childbearing potential
* Positive urine drug screen, except for lawfully prescribed medications and/or marijuana, provided that participant agrees to refrain from marijuana use during the period that they refrain from alcohol.
* Transaminases (AST or ALT) > 3.0 x the upper limit of normal
* Total bilirubin > 1.25 x the upper limit of normal
* Abnormal sodium, potassium, chloride, or bicarbonate levels that are considered potentially significant according to the clinical judgment of the PI.
* Creatinine equating to estimated glomerular filtration rate < 60 mL min-1 1.73 m-2
* Hemoglobin < 10 g/dL or hematocrit < 30%
* Platelet count < 100,000/μL
* Women currently pregnant, measured by serum and/or urine β-hCG
* Women currently breastfeeding
* History of having met any of the American Diabetes Association's definitions of prediabetic state during adulthood or diabetes mellitus (i.e., overt diabetes) at any time:

  * Hemoglobin A1c ≥ 5.7%, or rapid rise in documented HbA1c values causing clinical concern for evolving insulin deficiency
  * Plasma glucose ≥ 100 mg/dL after 8-h fast
  * Plasma glucose of ≥ 140 mg/dL at 2 h after ingestion of a 75-g glucose load
  * Random plasma glucose ≥ 200 mg/dL associated with typical hyperglycemic symptoms, diabetic ketoacidosis, or hyperglycemic-hyperosmolar state
* History of gestational diabetes mellitus within the previous 5 years
* Use of most antidiabetic medications within the 30 days prior to screening

  * Excluded: thiazolidinediones, sulfonylureas, meglitinides, DPP4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, amylin mimetics, acarbose, insulin
  * Metformin is acceptable provided that recruits meet all of the inclusion criteria at screening
* Known, documented history, at the time of screening, of any of the following medical conditions:

  * Pancreatic pathology, including but not limited to: Pancreatic neoplasia (unless appropriately evaluated and considered benign and not producing hormones), Chronic pancreatitis, History of acute pancreatitis within the past 5 years
  * Cardiovascular diseases (N.B. uncomplicated hypertension is not exclusionary)
  * Atherosclerotic cardiovascular disease
  * Stable or unstable angina
  * Myocardial infarction
  * Ischaemic or hemorrhagic stroke
  * Peripheral arterial disease (claudication)
  * Use of dual antiplatelet therapy (aspirin + P2Y12 inhibitor)
  * History of percutaneous coronary intervention
  * Heart rhythm abnormalities (non-sinus)
  * Congestive heart failure of any New York Heart Association class
  * Severe valvular heart disease (e.g., aortic stenosis)
  * Pulmonary hypertension
* Chronic kidney disease, Stage 3 or higher (estimated glomerular filtration rate < 60 mL/min/1.73 m2), of any cause
* Advanced or severe liver disease, including but not limited to:

  * Advanced liver fibrosis, as determined by non-invasive testing
  * Cirrhosis of any etiology
  * Autoimmune hepatitis or other rheumatologic disorder affecting the liver
  * Biliopathy (e.g., progressive sclerosing cholangitis, primary biliary cholangitis)
  * Hepatocellular carcinoma
  * Infiltrative disorders (e.g., sarcoidosis, hemochromatosis, Wilson disease)
* Gallstone disease, including:

  * Biliary colic (active)
  * History of acute cholecystitis not treated with cholecystectomy
  * History of other gallstone complications (e.g., pancreatitis, cholangitis)
* Chronic viral illness (N.B. diagnosis based only on medical history and not by laboratory confirmation)
* Hepatitis B virus (HBV), unless previously successfully eradicated with antiviral drugs that have been discontinued for at least 30 d prior to screening
* Hepatitis C virus (HCV) infection, unless previously successfully eradicated with antiviral drugs that have been discontinued for at least 30 d prior to screening
* Human immunodeficiency virus (HIV) infection
* Active seizure disorder (including controlled with antiepileptic drugs)
* Psychiatric diseases causing functional impairment that:

  * Are or have been decompensated within 1 year of screening, and/or
  * Require use of anti-dopaminergic antipsychotic drugs associated with significant weight gain/metabolic dysfunction (e.g., clozapine, olanzapine), monoamine oxidase inhibitors, tricyclic antidepressants, or lithium
* Other endocrinopathies:

  * Cushing syndrome (okay if considered in remission after treatment, provided that no exogenous corticosteroids or other ongoing treatment are required)
  * Adrenal insufficiency
  * Primary aldosteronism
* Venous thromboembolic disease (deep vein thrombosis or pulmonary embolism) or any required use of therapeutic anticoagulation
* Bleeding disorders, including due to anticoagulation, or significant anemia
* Active malignancy, or hormonally active benign neoplasm, except allowances for:

  * Non-melanoma skin cancer
  * Differentiated thyroid cancer (AJCC Stage I only)
* Clinical concern for increased risk of volume overload, including due to medications and/or heart/liver/kidney problems, as listed above
* Clinical concern for increased risk of hypokalemia, including low potassium on screening labs (i.e., below lower limit of normal), use of certain medications, or any medical conditions listed above
* Use of prescribed medications used for any of the indications in the preceding list of excluded conditions, or their use within 30 d prior to screening, except allowances for:

  * Use of drugs prescribed for indications other than the exclusionary diagnoses/purposes listed above (e.g., antiepileptic drugs used for non-seizure indications, ACEi/ARB used for uncomplicated hypertension rather than for congestive heart failure, etc.). Note, as above, that antidiabetic drugs except metformin within 30 d of screening are excluded.
* Oral or parenteral corticosteroids (at greater than prednisone 5 mg daily, or equivalent) for more than 3 days within the previous 30 days; topical and inhaled formulations are permitted.
* Beta blockers or non-dihydropyridine calcium channel blockers (verapamil or diltiazem)
* History of certain weight-loss (bariatric) surgery, including:

  * Roux-en-Y gastric bypass
  * Biliopancreatic diversion
  * Restrictive procedures (lap band, sleeve gastrectomy) performed within the past 6 months
* Clinical concern for alcohol overuse, including recent documented history during screening and/or participant report of regularly consuming more than 2 drinks per day for males or 1 drink per day for females.
* History of severe infection or ongoing febrile illness within 14 days of screening
* Any other disease, condition, or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
* Known allergy/hypersensitivity to any component of the medicinal product formulations, foods, IV infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
* Concurrent enrollment in another clinical study of any investigational drug therapy within 30 days prior to screening or within 5 half-lives of an investigational agent, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Steady-state plasma glucose at euinsulinemia (E-SSG) | 150-180 minutes during GIST protocol
  Plasma glucose level at steady state while insulin infusion rate is 4 mU/m2/min (units: mg/dL)
Steady-state plasma glucose at hyperinsulinemia (H-SSG) | 270-300 minutes during GIST protocol
  Plasma glucose level at steady state while insulin infusion rate is 32 mU/m2/min and glucose infusion rate is 267 mg/m2/min, reflective of insulin sensitivity (units: mg/dL)

SECONDARY OUTCOMES:
Steady-state plasma free fatty acids (FFA) at euinsulinemia | 150-180 minutes during GIST protocol
  Plasma FFA level while insulin infusion rate is 4 mU/m2/min (units: mmol/L)
Steady-state plasma free fatty acids (FFA) at hyperinsulinemia | 270-300 minutes during GIST protocol
  Plasma FFA level while insulin infusion rate is 32 mU/m2/min (units: mmol/L)

OTHER OUTCOMES:
Steady-state serum insulin at euinsulinemia (E-SSI) | 150-180 minutes during GIST protocol
  Serum insulin level at steady state while insulin infusion rate is 4 mU/m2/min (units: mU/L)
Steady-state serum insulin at hyperinsulinemia (H-SSI) | 270-300 minutes during GIST protocol
  Serum insulin level at steady state while insulin infusion rate is 32 mU/m2/min and glucose infusion rate is 267 mg/m2/min (units: mU/L)
Steady-state plasma glucagon level at euinsulinemia | 150-180 minutes during GIST protocol
  Plasma glucagon level while insulin infusion rate is 4 mU/m2/min (units: ng/L)
Steady-state plasma glucagon level at hyperinsulinemia | 270-300 minutes during GIST protocol
  Plasma glucagon level while insulin infusion rate is 32 mU/m2/min (units: ng/L)
Steady-state serum growth hormone (GH) level at euinsulinemia | 150-180 minutes during GIST protocol
  Serum GH level while insulin infusion rate is 4 mU/m2/min (units: ng/mL)
Steady-state serum growth hormone (GH) level at hyperinsulinemia | 270-300 minutes during GIST protocol
  Serum GH level while insulin infusion rate is 32 mU/m2/min (units: ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant-level clinical data will be preserved by depositing the deidentified data to Dryad, a generalist repository that is participating in the NIH Generalist Repository Ecosystem Initiative. The repository will provide metadata, persistent identifiers, and long-term access for open and controlled access. Each study created in Dryad is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication.
  To protect research participants' privacy and confidentiality, data submitted to the repository will not include personally identifiable information such as names or addresses. Additional protections, such as the approach for managing Health Insurance Portability and Accountability Act identifiers, will be used for de-identification and to provide a limited data set to minimize the risk of participant reidentification.
Time Frame: Scientific data will be shared as soon as possible. Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: To request access of the data, researchers will use the standard processes at Dryad. Given that we seek the widest possible availability, in most cases all that is necessary is obtaining a Dryad account from the repository web site.